CLINICAL TRIAL: NCT00135265
Title: Adolescent Smoking Cessation in Pediatric Primary Care
Brief Title: PROS Smokebusters: Adolescent Smoking Cessation in Pediatric Primary Care
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 15677
Record Dates: First submitted 2005-08-23; First posted 2005-08-25 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Health Care Quality, Access, and Evaluation; Smoking Cessation
Keywords: smoking cessation; adolescents
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Care Provider, Investigator

INTERVENTIONS:
Behavioral: smoking cessation, practice change — Providers will be trained in a brief smoking cessation intervention for teens.

SUMMARY:
This is a pilot study addressing office systems and clinician behavior change surrounding smoking cessation interventions for teens. The investigators' long-term goal is to improve the quality of clinical preventive services in practice-based research network settings. Their specific aims are to:

* a) pilot procedures for recruitment and randomization of PROS practices; and b) field trial/pilot PROS practitioner cessation counseling and practices' enrollment of adolescent patients; and
* assess the feasibility of pediatric clinician referral of adolescent patients to internet-based adjuncts for smoking cessation.

The investigators will evaluate a pilot round of recruitment and randomization, and smoking cessation training and delivery in 10 PROS practice sites; and assess the acceptability of study procedures and on-line internet counseling adjunct referral feasibility within PROS practice sites. Up to 1000 adolescents presenting for well visits will complete a short baseline survey prior to their well-visit. A sample of them will be surveyed by phone at 4-6 weeks to provide preliminary estimates of cessation counseling effectiveness for future studies. The investigators will field test measures, describe the patterns of smoking among youth, and explore how much receiving interventions affects motivation, quitting, abstinence/relapse attitudes, attitudes towards internet-based outreach strategies, and behaviors for 100 smokers.

**we have completed recruitment of providers; we are recruiting teens ONLY at this point**

DETAILED DESCRIPTION:
This is a pilot study addressing office systems and clinician behavior change surrounding smoking cessation interventions for teens. The investigators' long-term goal is to improve the quality of clinical preventive services in practice-based research network settings. Their specific aims are to:

* a) pilot procedures for recruitment and randomization of PROS practices; and b) field trial/pilot PROS practitioner cessation counseling and practices' enrollment of adolescent patients; and
* assess the feasibility of pediatric clinician referral of adolescent patients to internet-based adjuncts for smoking cessation.

The investigators will evaluate a pilot round of recruitment and randomization, and smoking cessation training and delivery in 10 PROS practice sites; and assess the acceptability of study procedures and on-line internet counseling adjunct referral feasibility within PROS practice sites. Up to 1000 adolescents presenting for well visits will complete a short baseline survey prior to their well-visit. A sample of them will be surveyed by phone at 4-6 weeks to provide preliminary estimates of cessation counseling for future studies. The investigators will field test measures, describe the patterns of smoking among youth, and explore how much receiving interventions affects motivation, quitting, abstinence/relapse attitudes, attitudes towards internet-based outreach strategies, and behaviors for 100 smokers.

ELIGIBILITY:
Inclusion Criteria:

Practitioner recruitment criteria:

* Has a patient flow of several adolescents per week.
* Reads and speaks English.
* Able and willing to provide informed consent

Patient recruitment criteria:

* 14 years or older
* Lives in a home or apartment with access to a phone or mail address
* Speaks English
* Cognitively able to respond to survey questions
* Cognitively able to give assent and obtain parent/guardian permission or consent

Exclusion Criteria:

* Providers: already participating in a PROS study

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4100 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
smoking cessation rates | 4-6 weeks
quit attempts | 4-6 weeks
provider practice change | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan D Klein, MD, MPH, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States